CLINICAL TRIAL: NCT05123248
Title: Integrating the Use of Calibration-Free Continuous Monitoring for Pregnancy Glucose Profiling: I-Profile Study
Acronym: I-Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/2128
Record Dates: First submitted 2021-10-25; First posted 2021-11-17 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Gestational Diabetes; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Participants randomized to both the non-blinded continous glucose monitoring sensors and the blinded continous glucose monitoring sensors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Blinded Group (Experimental): Participants in the blinded group will be wearing the sensor for 14 days without a reader. After 14 days, participants are required to scan the sensor themselves or with the assistance of a CRC to a designated blinded-reader.
  Interventions: Device: Blinded Group
- Unblinded Group (Experimental): Participants in the non-blinded group are required to wear the sensor for 14 days with an open reader. The participant will be required to upload their glucose readings no longer than 8 hours by scanning the reader provided.
  Interventions: Device: Unblinded group

INTERVENTIONS:
Device: Blinded Group — Participants in the blinded group will be wearing the sensor for 14 days without a reader. Glucose levels will be recorded from the interstitial fluid every 15 minutes using intermittent/ flash glucose scanning. After 14 days, participants are required to scan the sensor themselves or with the assistance of a CRC to a designated blinded-reader.
  Arms: Blinded Group
Device: Unblinded group — Participants in the non-blinded group are required to wear the CGM sensor for 14 days with an open reader. Glucose levels will be recorded from the interstitial fluid every 15 minutes using intermittent/ flash glucose scanning. The participant will be required to upload their glucose readings no longer than 8 hours by scanning the reader provided.
  Arms: Unblinded Group

SUMMARY:
This study aims to test the following hypotheses in a longitudinal, observational study in pregnant women who will be randomized to received either a Blinded or Unblinded CGM sensor and followed-up 6-12 weeks after delivery:

1. CF-CGM device is well tolerable and accurate for glucose level monitoring in women with a normal pregnancy.
2. CF-CGM device is well tolerable and acceptable in women with GDM who are required intensive glucose monitoring on a daily basis during pregnancy and even after delivery.
3. There are trimester-specific glucose profiles observed in the whole pregnancy.
4. Pregnancies complicated with GDM would show a specific glucose profile that is different from non-GDM pregnancies (e.g. greater daily fluctuations, more episodes and longer duration of glucose spikes after meal).
5. There is a good correlation between one-day glucose profile and OGTT test at 24-31 weeks gestation GDM screening.
6. Pre-GDM screening glucose profiles is predictive of GDM diagnosis at 24-31 weeks gestation.

DETAILED DESCRIPTION:
GDM affects 5-10% of pregnant women in Europe, while the prevalence in Asian populations is significantly higher at approximately 15-20%. However, the GDM screening approaches, timing and targeted population still varies greatly in clinical practice all over the world, which makes the prevalence of GDM difficult to compare universally. Since the early days of the 21st century, the continuous glucose monitoring system (CGM) has been used for constant evaluation of glucose levels by measuring interstitial glucose concentrations. It can potentially improve diabetes care if used carefully with proper understanding of the characteristics of this system.

This is longitudinal, observational and hospital-based study. A total of 500 pregnant women will be recruited with consent form completion after meeting our inclusion criteria. The recruited women will then be randomly assigned to a Blinded and Unblinded CGM device.

All pregnant women aged 21 and above who plan to be followed up throughout pregnancy and intend to deliver at KKH and currently attending KKH for antenatal consultation during their early trimester will be approached by study research personnel, and will be followed up from then onwards. If they agree to take part in the study, consent will be signed at the first trimester clinic visit.

All recruited subjects will be randomized to put on a Blinded or Unblinded CGM device for 14 days from the first trimester (9-13 weeks), 18-23 weeks, 24-31 weeks, and 32-33 weeks. If a pregnant subject is diagnosed with GDM using International association of diabetes and pregnancy study groups (IADPSG) guidelines at KKH at 24-31 weeks gestation, she will be required to wear the sensor continuously until 38 weeks gestation, and will be followed up for another 14 days at the 6-12 weeks postnatal period.

Data will be collected through questionnaires and clinical measurements. The questionnaires include socio-economic factors, medical histories, lifestyle factors, health status, and home environment. Bio-physical measurements will be obtained from anthropometric measurements of participants, human biological materials such as blood, are collected from the participants at their follow-up time points with the I-PROFILE study upon their consent.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are Singapore citizens or Singapore Permanent Residents, and plan to be followed up throughout pregnancy and intend to deliver at KKH;
2. Aged 21 and above;
3. Singleton pregnancy

Exclusion Criteria:

1. Have serious skin conditions (e.g. eczema) that precludes wearing the sensor for 14 days;
2. Patients who have any other chronic disease such as chronic kidney disease.
3. Unable to read or speak English

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Gestational Diabetes Mellitus (GDM) | 24-31 weeks gestation
  Clinical outcomes of Gestational Diabetes Mellitus (GDM) development determined by oral glucose tolerance test

SECONDARY OUTCOMES:
CGM summary metrics derived from extracted CGM glucose data | First trimester: 9-13 weeks, Second trimester: 18-23 weeks, 24-31 weeks, 32-33 weeks
  Glucose profiles extracted from the continous glucose monitoring (CGM) device
Plasma glucose measures from OGTT | 24-31 weeks gestation
  Fasting, one hour and 2 hour glucose values obtained from OGTT

OTHER OUTCOMES:
Applicability, acceptability, compliance of the blinded the CGM device use in a normal pregnancy. | At 32-33 weeks gestation
  Using a 10-item patient feedback survey
Applicability, acceptability, compliance of the unblinded the CGM device use in a normal pregnancy. | At 32-33 weeks gestation
  Using a 14-item patient feedback survey
Applicability, acceptability, compliance of the blinded CGM device use in a GDM pregnancy | 6-12 weeks postnatal
  Using 10-item patient feedback survey
Applicability, acceptability, compliance of the unblinded CGM device use in a GDM pregnancy | 6-12 weeks postnatal
  Using a 14-item patient feedback survey

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quah PL, Tan LK, Thain SPT, Lek N, Tagore S, Chern BSM, Ang SB, Wright A, Jong M, Tan KH. First Trimester Mean Glucose Level on Continuous Glucose Monitoring Is Associated with Infant Birth Weight. Diabetes Metab J. 2025 Nov;49(6):1262-1271. doi: 10.4093/dmj.2024.0700. Epub 2025 Jun 2. PMID 40452210